CLINICAL TRIAL: NCT05804409
Title: Screening for Pancreatic Exocrine Insufficieny in Metabolic Associated Fatty Liver Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Ahmed Mahmoud Hammam, Ghada Ahmed Mahmoud Hammam, Assiut University
Other Study IDs: PEI in MAFLD
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Exocrine Insufficiency
Keywords: MAFLD
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FECAL ELASTASE — screening for pancreatic exocrine insufficiency in MAFLD patients

SUMMARY:
to investigate the frequency of PEI in MAFLD

DETAILED DESCRIPTION:
The growing epidemic of obesity is observed worldwide as lifestyles change to include higher caloric diets and decreasing physical activity.

With obesity; ectopic fat deposition in certain organs is accompanied by insulin resistance, hypertension and dyslipidemia; which in turn leads to metabolic syndrome As such, metabolic associated fatty liver disease (MAFLD), the hepatic manifestation of metabolic syndrome, has already become the most common cause of liver disease worldwide with a prevalence 25% Another important organ where ectopic fat deposition takes place is pancreas. Although hepatic fat is mainly intracellular and fatty pancreas is a consequence of adipocyte infiltration, evidence exists that fatty pancreas could be used as the initial indicator of ectopic fat deposition Recently, an advanced MRI technique - MRI-estimated proton density fat fraction (MRI-PDFF) - was shown to give reliable quantitative information of hepatic fat that is well correlated with liver biopsy The pancreas is composed of two glands - endocrine pancreas and exocrine pancreas- that are intimately mixed together into one organ Although exocrine pancreas comprise more than 95% of the pancreatic mass, to date there is no study conducted about the exocrine pancreas function and pancreatic fat in MAFLD patients The fecal pancreatic elastase (PE) test is a valuable indirect assay used in the evaluation of pancreatic exocrine function PE testing has become a standard diagnostic tool exhibiting good correlation with the results of direct functional tests as well as morphological changes in the pancreas discovered via imaging techniques In the last decade, significant number of studies were conducted on pancreatic exocrine insufficiency (PEI)

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years, Patients diagnosed as MAFLD

Exclusion Criteria:

* Patients use steatogenic medications, hormone replacement therapy or herbal products, any alcohol intake.

  * Patients with any history of pancreatic diseases like acute pancreatitis, chronic pancreatitis and pancreatic surgery.
  * Patients with any malignancy.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: MAFLD is diagnosed in patients when they have both hepatic steatosis and any of the following three metabolic conditions: overweight/obesity, diabetes mellitus, or evidence of metabolic dysregulation (MD) in lean individuals.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
investigate the frequency of PEI in MAFLD | baseline
  screening for PEI by fecal elastase test in MAFLD patients

REFERENCES:
- [Background] Boga S, Koksal AR, Sen I, Kurul Yeniay M, Yilmaz Ozguven MB, Serin E, Erturk SM, Alkim H, Alkim C. Liver and pancreas: 'Castor and Pollux' regarding the relationship between hepatic steatosis and pancreas exocrine insufficiency. Pancreatology. 2020 Jul;20(5):880-886. doi: 10.1016/j.pan.2020.04.020. Epub 2020 May 19. PMID 32475757
- See also: screening for PEI in MAFLD patients — https://doi.org/10.1016/j.pan.2020.04.020